CLINICAL TRIAL: NCT01187589
Title: Preliminary Assessment of the Effect of PulseHaler™ With Albuterol on Lung Deposition of Aerosol and on Pulmonary Functions in COPD Patients
Brief Title: PulseHaler Drug Deposition Study in Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Respinova LTD (Industry)
Responsible Party: Yuval Avni, Respinova LTD
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PLS-02
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulsehaler (Experimental): Fully operational Pulsehaler, with protocol enabled
  Interventions: Device: Pulsehaler; Drug: Nebulizer & Albuterol 0.5ml
- Nebulizer (Active Comparator): Deactivated Pulsehaler (protocol disabled), so only the nebulizer is active
  Interventions: Drug: Nebulizer & Albuterol 0.5ml

INTERVENTIONS:
Device: Pulsehaler
  Arms: Pulsehaler
Drug: Nebulizer & Albuterol 0.5ml — Albuterol aerosolized by a nebulizer

SUMMARY:
This study is aimed at finding the effect of PulseHaler™ with Albuterol on Lung Deposition of Aerosol and on Pulmonary Functions in COPD Patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD), established for at least 1 year
* Post-bronchodilator FEV1/FVC < 0.7
* Post-bronchodilator FEV1 in the range 30% - 70% predicted
* Age: 40 years or older
* Patient signed the informed consent form

Exclusion Criteria:

* Pneumothorax in the past, per anamnesis.
* Women at the age of fertility, who are pregnant, or plan pregnancy, or do not use contraceptive.
* Severe cardiac disease, e.g., Congestive Heart Failure (CHF) grade 3 or higher
* Coronary Artery Bypass Graft (CABG) or Acute Myocardial Infarction (MI) within last 3 months
* Other severe systemic disease
* Non-cooperative or non-compliant patient

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Lung deposition | 1 hour
  Lung deposition of the albuterol-containing aerosol
Pulmonary functions | 1 hour
  Pulmonary function tests by spirometry

SECONDARY OUTCOMES:
Dyspnea | 1 hour
  Dyspnea measured by the modified Borg scale

CONTACTS AND LOCATIONS:
Overall Officials: Haim Golan, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center Nuclear Medicine Institute, Tzrifin, Israel